CLINICAL TRIAL: NCT06164366
Title: Patient Satisfaction and Adaptation of Maxillary Resin Dentures Printed at 0 Versus 45 Degrees Build Angle: A Randomized Pilot Cross-over Clinical Trial
Brief Title: Patient Satisfaction and Adaptation of Dentures Printed at 0 Versus 45 Degrees
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Iman Abd-ElWahab Radi, PhD, Professor, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 245326677
Record Dates: First submitted 2023-08-06; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Edentulous Jaw
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0 Degrees Group (Experimental): dentures will be printed at a 0 degrees build angle
  Interventions: Device: 0 degrees 3D printed upper complete dentures
- 45 Degrees Group (Active Comparator): dentures will be printed at a 45 degrees build angle
  Interventions: Device: 45 degrees 3D printed upper complete dentures

INTERVENTIONS:
Device: 0 degrees 3D printed upper complete dentures — 3d printed dentures at a build angle of 0 degrees
  Arms: 0 Degrees Group
Device: 45 degrees 3D printed upper complete dentures — 3d printed dentures at a build angle of 45 degrees
  Arms: 45 Degrees Group

SUMMARY:
This pilot study aims to compare the difference, if present in patient satisfaction, denture base adaptation and retention in 3d printed maxillary complete dentures fabricated at a build angle of 0 degrees versus 45 degrees.

DETAILED DESCRIPTION:
This pilot study aims to compare the difference, if present in patient satisfaction, denture base adaptation and retention in 3d printed maxillary complete dentures fabricated at a build angle of zero degrees versus forty five degrees. Since there is no sufficient evidence surrounding the topic at hand, a randomized clinical trial must be conducted in an attempt to gap the clinical knowledge regarding printing orientation and its effect on denture base adaptation and patient satisfaction. The main question and the one that needs further investigations as stated by Goodacre would these differences in these build up angles have a true clinical effect on denture adaptation and denture retention

ELIGIBILITY:
Inclusion Criteria:

1. Patients above the age of 40
2. Patients with opposing full natural dentition or completely or partially edentulous arches
3. Opposing arch should be either having a set of full natural dentition or is restored by fixed partial dentures or implants
4. Cooperative patients that are willing to attend all follow-up periods.
5. Patients with healthy attached mucosa of appropriate thickness free from any inflammation.

6- Patients free from any systemic disease that might affect the health of the bone or of the mucosa eg diabetes

Exclusion Criteria:

1. Patients with any temporomandibular joint disorder or parafunctional habits
2. Patients with flabby or flat ridges
3. Patients with extreme anatomical limitations such as a large torus that requires surgical excision.
4. Patients with a history of allergy to dentures made of resins.
5. Patients with pathological changes of residual ridges as recurrent or persistent ulcers, osteomyelitis and infections.
6. Patients with medical or psychological conditions as physical disability or mental retardation that hinder cooperation in the follow up visits and answering the questionnaires.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
patient satisfaction | 6 months
  Measured through a questionnaire using a likert scale from 1 - 5 with 1 being extremely satisfied with the intervention and 5 being extremely satisfied with the intervention
denture adaptation | 4 weeks
  measured using 3d metrology software in terms of the root mean square (RMS) values of trueness and adaptation

SECONDARY OUTCOMES:
Denture retention | 6 months
  Measured using Kapur scoring system. The grading will follow a Scoring System with four possible scores for retention from least (0) to best retention (3)

IPD SHARING:
Plan to Share IPD: No